CLINICAL TRIAL: NCT00480012
Title: The Effects of Transcranial Magnetic Stimulation of the Brain on Memory-consolidation in Human Primary Visual Cortex
Brief Title: The Effects of TMS on Memory-consolidation in Human Primary Visual Cortex
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to administrative issues, the study was withdrawn.
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Amiaz Revital, MD - Senior Psychiatrist, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SHEBA-04-3437-RA-CTIL
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: healthy subjects

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Device: rTMS — repetitive transcranial meagnetic stimulation of the brain

SUMMARY:
Rapid Transcranial Magnetic Stimulation will be used in order to examine whether the human primary visual cortex is essential to visual memory consolidation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Right handed

Exclusion Criteria:

* Active/past neurological/psychiatric disorder
* Personal/first-degree history of seizures
* Cardio-vascular disorder or disease including hypertension chronic use of medication
* Metal/electronic device implant
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Estimated)
Dates: Start 2005-05; Primary Completion 2007-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Revital Amiaz, MD, Principal Investigator — Sheba Medical Center